CLINICAL TRIAL: NCT02539732
Title: Prediction of Outcome of Weaning From Mechanical Ventilation Using the Electrical Activity of the Diaphragm
Acronym: OWED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: REB# 15-214
Record Dates: First submitted 2015-08-27; First posted 2015-09-03 (Estimated); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Respiratory Insufficiency
Keywords: Weaning; Spontaneous breathing trial; Neurally-adjusted ventilator assist; Electrical activity of the diaphragm
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Several types of spontaneous breathing trials (SBTs) have been proposed to evaluate when a patient is ready to be weaned from the ventilator based on breathing pattern measurements. The T-piece technique allows clinicians to calculate breathing patterns accurately but many prefer to use minimal levels of assistance, which unfortunately modifies breathing pattern. The interest of Neurally Adjusted Ventilatory Assist (NAVA) is that tidal volume (Vt) supposedly represents what the patient really wants: without disconnecting the patient from the ventilator, it may be possible to determine what is the real need and whether the patient is able to maintain Vt without support. The aims of the study are as follows: to test whether the changes in Vt after the removal of a standardized level of NAVA assistance (ΔVt) can predict weaning outcome; to compare the proposed titration of effort in NAVA (occlusion) with Patient-Ventilator Breath Contribution (PVBC) and titration using the Pmusc/Eadi index (PEI) relating the pressure generated by the respiratory muscles (muscular pressure; Pmusc) to the electrical activity of the diaphragm (EAdi); to assess the effect of PEEP on the change in Vt; and to evaluate EAdi after extubation. Patients ventilated for at least 24 hours who are ready to undergo an SBT will be included. Patients younger than 18 years of age and/or who have a contraindication to NAVA catheter insertion and/or surgical patients expected to be extubated within 12 hours will be excluded. After a baseline inclusion period with the pre-enrollment mode of ventilation, the standardized NAVA level will be applied for 20 minutes, during which both Patient-Ventilator Breath Contribution (PVBC) and PEI will be calculated. After the NAVA trial, a period of Continuous Positive Airway Pressure (CPAP) 5 (2-3 minutes) followed by a period of CPAP 0 (2-3 minutes) (both with NAVA gain 0) will be performed in order to record the difference with Vt during standardized NAVA (ΔVt). At the end of this period, the patient will be switched back to the baseline settings for 30 minutes-3 hours. After this period, the patient will perform an SBT with CPAP 0 or CPAP 5 for 1 hour. At the end of the SBT, the attending physician will decide whether or not to extubate the patient according to standard criteria and blinded to the ΔVt results. Ultimately, patients will be classified as "success" or "failure" and the ΔVt will be compared between these two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients ready to undergo an SBT based on the decision of the clinical team.
* Patients ventilated for at least 24 hours

Exclusion Criteria:

* Patients younger than 18 years-old
* Contraindication to NAVA catheter insertion (e.g., recent surgery, bleeding)
* Central Neurological disorder (hemorrhage, tumor, massive stroke, etc.) heavily influencing breathing pattern
* Surgical patients expected to be extubated within 12 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated Intensive Care Unit patients who are ready to undergo a Spontaneous Breathing Trial.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2015-09; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in tidal volume after removing a standardized level of NAVA assistance. | Up to 3 hours

SECONDARY OUTCOMES:
Comparison of Pmusc estimated by an occlusion technique, PVBC, and PEI. | Up to 3 hours
Change in tidal volume from PEEP of 5 centimeters of water (cmH2O) to zero PEEP. | Up to 3 hours
Change in EAdi during NAVA mode, CPAP, and after extubation. | Up to 7 days

CONTACTS AND LOCATIONS:
Locations (3):
- St. Michael's Hospital, Toronto, Ontario, Canada
- Centre Hospitalier Universitaire Angers, Angers, France
- Azienda Ospedaliero - Universitaria OORR Ospedali Riuniti di Foggia, Foggia, Italy

REFERENCES:
- [Background] Yang KL, Tobin MJ. A prospective study of indexes predicting the outcome of trials of weaning from mechanical ventilation. N Engl J Med. 1991 May 23;324(21):1445-50. doi: 10.1056/NEJM199105233242101. PMID 2023603
- [Background] Bellani G, Mauri T, Coppadoro A, Grasselli G, Patroniti N, Spadaro S, Sala V, Foti G, Pesenti A. Estimation of patient's inspiratory effort from the electrical activity of the diaphragm. Crit Care Med. 2013 Jun;41(6):1483-91. doi: 10.1097/CCM.0b013e31827caba0. PMID 23478659